CLINICAL TRIAL: NCT05744739
Title: Phase 1 Dose Escalation Study of Tomivosertib in Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Tomivosertib in Relapsed or Refractory Acute Myeloid Leukemia (AML)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); EFFECTOR Therapeutics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 22H08; NCI-2023-00767 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NU 22H08; STU00218776 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; tomivosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (tomivosertib) (Experimental): Tomivosertib will be dosed continuously on days 1-28 of each 28-day cycle.
  Interventions: Procedure: Biospecimen Collection; Drug: Tomivosertib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Tomivosertib — Given PO
  Other Names: EFT-508; eFT508; Spiro(cyclohexane-1,3'(2'H)-imidazo(1,5-a)pyridine)-1',5'-dione, 6'-((6-Amino-4-pyrimidinyl)amino)-8'-methyl-

SUMMARY:
Phase 1 of the study will open first with a (Bayesian optimal interval BOIN) dose finding design. The starting dose of tomivosertib is 100mgdaily (doses 24 ± 2 hours apart), PO, self-administered with meals. The dose finding follows a BOIN design, with the 100mg BID dose level with a meal being the highest dose. There is one dose level below (dose level -1 = 100mg QD without a meal) that will be given if the de-escalation condition is met during dose finding. Upon completion of the phase 1 dose finding portion of the study, the recommended starting dose of tomivosertib for the subsequent combination with the other agents will be determined, as described in Section 4.3 and Section 8.0.

Tomivosertib will be dosed continuously on days 1-28 of each 28-day cycle at the dose level assigned for that cohort.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To determine the dose of maximum pharmacologic activity (MPA) of tomivosertib in relapsed/refractory AML .

SECONDARY OBJECTIVES:

1. To assess the adverse event profile of tomivosertib
2. To estimate the rate of complete remission (CR)
3. To estimate the rate of overall response
4. To estimate the duration of response (DOR)
5. To estimate progression free survival (PFS)
6. To estimate overall survival (OS)
7. To assess the outcomes for patients who undergo allogeneic hematopoietic stem cell transplant (HSCT)
8. To assess the pharmacodynamics of tomivosertib by eIF4E phosphorylation before, during, and after cycle 1 treatment
9. To measure MCL1 expression before and after cycle 1 treatment
10. To assess the steady-state pharmacokinetics of tomivosertib

EXPLORATORY OBJECTIVES:

1. To correlate eIF4E phosphorylation before and after cycle 1 treatment with treatment response.
2. To correlate MCL1 expression before and after treatment with treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >= 18 years
* Patients with relapsed/refractory AML (based on the International Consensus Classification of Myeloid Neoplasms and Acute Leukemias

Previous treatment must consist of:

1. At least 1 cycle of therapy with an anthracycline and standard dose cytarabine containing regimen; OR
2. At least one cycle of a high- or intermediate-dose cytarabine containing regimen; OR
3. At least 4 cycles of hypomethylating agent (HMA) as single agent or 2 cycles of HMA and venetoclax; OR
4. Allogeneic stem cell transplant (SCT) for either AML or high-risk MDS and have recovered from all transplant-related toxicities, are off all immunosuppression for at least 6 weeks, and have no evidence of acute or chronic graft-versus-host disease GvHD); OR
5. Relapsed or refractory disease without established alternative therapy.

   * For patients with a known history of human immunodeficiency virus (HIV), infected patients on effective anti-retroviral therapy must have a viral load undetectable for 6 months prior to registration.
   * For patients with a known history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
   * Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
   * Patients must agree to serial bone marrow aspirate/biopsies
   * The effects of tomivosertib on the developing human fetus are unknown. For these reasons, patients of child-bearing potential (POCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) and refrain from donating eggs from the time of informed consent, for the duration of study treatment, and for 30 days following completion of study therapy. Should a patient become pregnant or suspect they are pregnant while they or their partner are participating in this study, they should inform their treating physician immediately.

People with sperm-producing reproductive capacity treated or enrolled on this protocol must also agree to use adequate contraception (or abstinence or vasectomy) and refrain from donating sperm from the time of informed consent, for the duration of study therapy, and 30 days after completion of study therapy.

NOTE: A POCBP is any person with an egg-producing reproductive tract (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy
* Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* POCBP (defined in 3.1.7) must have a negative serum β-subunit of human chorionic gonadotropin (β-hCG) pregnancy test (sensitivity of at least 25 mIU/mL) within 14 days prior to registration on study and have a negative serum β-hCG pregnancy test (sensitivity of at least 25 mIU/mL) within 72 hours prior to the start of study treatment.

NOTE: The screening serum pregnancy test can be used as the test prior to the start of study treatment if it is performed within the 72-hour timeframe.

- Patients must provide written, signed, and dated informed consent prior to study registration. Patient must have the ability to understand and the willingness to sign a written informed consent document. The patient must be willing and able to comply with the protocol for the duration of the study. NOTE: No study-specific screening procedures may be performed until written consent has been obtained

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* Previous chemotherapy including biologic/targeted therapy or immunological agents for AML within 14 days prior to start of tomivosertib..
* Patients who have a prior or concurrent malignancy that may interfere with study treatment or safety. NOTE: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen (i.e., cancers under observation that do not require treatment, resectable skin cancer, low risk prostate cancer, DCIS, LCIS, etc.) are eligible per lead PI discretion. Patients with prior MDS or MPN are eligible.
* Patients who have conditions that would interfere with drug absorption
* Patients who have conditions that would interfere with their ability to swallow oral medications
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to tomivosertib, azacitidine, and/or venetoclax
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Uncontrolled systemic infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, antifungal therapy and/or other treatment)
  * Unstable angina pectoris
  * Cardiac ventricular arrhythmia, except for patients that can be successfully treated with rate control or anti-arrhythmic agents
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Patients who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2030-04-23 (Estimated)

PRIMARY OUTCOMES:
Determine the dose of maximum pharmacologic activity (MPA) of tomivosertib | From the initiation of trial therapy (cycle 1 day 1), and throughout the first cycle of treatment for a total of 28 days
  The 'MPA' is defined as the minimum dose of tomivosertib tested in the phase 1 dose-finding portion of the trial that the isotonic estimate of dose-limiting toxicities (DLTs) is below or equal to the target DLT rate of 20% in phase 1 and biologic activity is observed. Whichever dose level is declared the MPA must have at least 6 patients treated at that level.

SECONDARY OUTCOMES:
Frequency of adverse events | Up to 18 months
  Safety and tolerability will be summarized by providing a frequency of adverse events (CTCAE version 5.0) by severity, type, timing, and attribution for toxicities of any grade, with rates of >= grade 3 toxicities also analyzed separately. Adverse event rates will be summarized and accompanied by 95% exact binomial confidence intervals.
Overall response rate | Up to 18 months
  The proportion of treated patients who experience an objective response (complete remission [CR], complete remission with incomplete platelet recovery [CRp], complete remission with incomplete hematological recovery [CRi] and partial remission [PR]) per International Working Group AML Response Criteria. Will be summarized as a proportion with a corresponding exact 95% confidence interval (CI).
Complete remission rate (CRR) | Up to 18 months
  The proportion of treated patients who experience CR, CRp, and CRi will be reported. The first date of response for CR, CRp, or CRi will be used for the calculation of CRR. Will be summarized as a proportion with a corresponding exact 95% CI.
Duration of response (DOR) | Time between the day of first documented response to trial therapy (CR, CRp, and CRi or PR), whichever is first recorded, and subsequent disease progression, assessed up to 18 months
  Will be analyzed using the Kaplan-Meier method. The median of DOR, if estimable, will be reported along with the confidence intervals.
Progression free survival (PFS) | Time between the initiation of trial therapy and the day of first documented disease progression or death from any cause, assessed up to 18 months
  Will be analyzed using the Kaplan-Meier method. The median of PFS, if estimable, will be reported along with the confidence intervals.
Overall survival (OS) | Time between the initiation of trial therapy and the date of death from any cause, assessed up to 18 months
  Will be analyzed using the Kaplan-Meier method. The median of OS, if estimable, will be reported along with the confidence intervals.
To assess the pharmacodynamics of tomivosertib by eIF4E phosphorylation before, during, and after cycle 1 treatment | Baseline and after Cycle 1 treatment
  Phosphorylation of eIF4E will be assessed by flow cytometry in order to identify a biologically effective dose.
OS for patients who proceed to transplant | From initiation of therapy until the patient completes follow-up, or experiences death from any cause, assessed up to 18 months
  Will estimate the OS for patients who proceed to transplant, compared to those who do not undergo transplant.

OTHER OUTCOMES:
Measure MCL1 expression before and after cycle 1 treatment | Baseline and after Cycle 1 treatment
  Using flow cytometry, the correlation between decreased MCL1 expression after treatment and favorable response to treatment will be determined.
Assess the steady-state pharmacokinetics of tomivosertib | Up to 18 months
  PK analysis will be done using the PK population
Correlate eIF4E phosphorylation before and after cycle 1 treatment with treatment response. | Baseline and after Cycle 1 treatment
  correlation between high Correlation of phosphorylation levels of eIF4E at baseline and favorable response to treatment
Correlate MCL1 expression before and after treatment with treatment response. | Baseline and after Cycle 1 treatment
  Using flow cytometry, view the correlation between decreased MCL1 expression after treatment and favorable response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shira N Dinner, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States